CLINICAL TRIAL: NCT04693000
Title: Use of Topical Solasodine of Solanum Melongena Peel Origin in the Treatment of Palmar Arsenic Keratosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr Mohammad Sazzad Hossain, MBBS, MD(Phase B) Resident, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BSMMU/2019/10655
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Keratotic Nodular Size
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Keratosis lesion or nodular size observation after 12 weeks of therapy with solasodine ointment (Experimental): An ointment containing solasodine extract of solanum melongena peel origin applied to patients with palmar arsenical keratosis; dose-twice daily for 12 weeks.
  Keratotic nodular size observation after 12 weeks
  Interventions: Drug: Arsenic Keratosis lesion or nodular size observation after 12 weeks of therapy with solasodine ointment

INTERVENTIONS:
Drug: Arsenic Keratosis lesion or nodular size observation after 12 weeks of therapy with solasodine ointment — An ointment containing solasodine extract of solanum melongena peel origin applied to patients with palmar arsenical keratosis; dose-twice daily for 12 weeks.Keratotic nodular size observation after 12 weeks

SUMMARY:
Arsenic is one of the largest mass poisonings in Bangladesh. Arsenic keratosis of the palm and sole is a common feature of arsenicosis. Brinjal or eggplant ubiquitous vegetable found in different parts of the world, including Bangladesh, scientifically known as Solanum melongena. A study showed ointment containing crude extract of Solanum melongena peel origin is effective in arsenic keratosis. Solasodine is one of the active compounds of Solanum melongena peel. In the current study, an ointment containing a single compound solasodine isolated from Solanum melongena peel . The ointment made from solasodine extract was distributed among arsenic keratosis patients to see the effect.

DETAILED DESCRIPTION:
About millions of Bangladeshi people are chronically exposed to high arsenic concentrations (above 50 micrograms/liter) through contaminated drinking water and thus suffer from arsenic-related health hazards called arsenicosis. Arsenic keratosis is one of the commonest skin manifestations of arsenicosis that occur in the palm and sole that is troublesome for the working people and females suffered a negative socio-economic impact.

Two studies were conducted in the same department where topical ointment prepared from the crude extract of S. melongena peel was found effective in arsenical keratosis.

The present study was conducted to confirm the previous study and identify that solasodine isolated from S. melongena peel is responsible for the cure of the lesions of arsenical keratosis. Thus, it may be possible for the chemical synthesis of solasodine, and an effective, inexpensive topical ointment can be prepared for the cure of arsenical keratosis.

ELIGIBILITY:
Inclusion Criteria:

* Presence of moderate to severe palmar arsenical keratosis
* Drinking arsenic-contaminated water for at least six months
* Patient voluntarily agreed to participate

Exclusion Criteria:

* Age less than 18 years or more than 60 years
* Pregnant and nursing mother
* Skin diseases like atopic dermatitis eczema and psoriasis
* Patient allergic to brinjal (eggplant)
* Patient taken any treatment of arsenicosis for the last six months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-23 (Actual); Primary Completion 2021-01-15 (Estimated); Study Completion 2021-01-15 (Estimated)

PRIMARY OUTCOMES:
Arsenical Keratotic nodular size of the palm | 12 weeks
  Keratotic nodular size or lesion size will be measured by slide calipers

CONTACTS AND LOCATIONS:
Locations (1):
- Muradnagar Upazilla, Comilla, Bangladesh

IPD SHARING:
Plan to Share IPD: No